CLINICAL TRIAL: NCT00060983
Title: Effects of Sensory Motor Input on Gait in SCI (Spinal Cord Injured) Subjects
Brief Title: Improving Gait in Patients With Spinal Cord Injuries
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5K01HD001193-02 (NIH)
Record Dates: First submitted 2003-05-16; First posted 2003-05-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-05

CONDITIONS: Spinal Cord Injuries
Keywords: Locomotion; Spinal Cord Injury, ASIA C; Body weight support (BWS); Functional electrical stimulation (FES); Gait; Treadmill training; Physical Therapy
MeSH Terms: conditions — Spinal Cord Injuries

INTERVENTIONS:
Procedure: Body weight supported locomotor training
Procedure: Functional electrical stimulation

SUMMARY:
This study is part of a larger clinical trial that examines the potential of a 12-week treadmill-training program to improve walking in patients with spinal cord injuries (SCIs). Patients in the trial are at least 1 year past their injury. This substudy tests a combination of two strategies to enhance the treadmill training program: electrically stimulating a muscle withdrawal reflex and providing body weight support by partially suspending patients as they walk on the treadmill.

DETAILED DESCRIPTION:
Patients with spastic paresis due to incomplete SCI have inadequate motor control of the lower extremities that results in a number of abnormalities of movement. Among these are unregulated spinal reflexes, inadequate and delayed motor recruitment, and balance deficits. If the patient can walk, these abnormalities manifest in a gait pattern that has poorly coordinated timing between different muscle groups, decreased weight bearing capacity, and inappropriate muscle activity, such as scissoring.

Research in patients with SCIs has demonstrated that, despite the damage to the spinal cord, many of the nervous system pathways that control walking remain intact and can be activated by the proper sensory stimulation. Two technologies that may enhance the benefits of treadmill walking are body weight support (BWS) and functional electrical stimulation (FES). Preliminary studies indicate that by combining these two interventions, gait performance is improved such that more efficient and functional movement emerges. This study will evaluate the benefits of adding BWS and FES to a treadmill-training program for patients with SCIs.

During the treadmill training, patients are suspended in an apparatus to provide partial body weight support (BWS). The training effects of BWS locomotion with FES over the course of a multi-session training program will be examined. Study visits will be scheduled 3 days each week for 12 weeks. Participants will have follow-up visits at Months 3 and 12. Gait parameters modified by training will be identified and the nature of these changes will be characterized. Specifically, walking speed, kinematics, electromyography (EMG), and muscle strength will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury classified as American Spinal Injury Association (ASIA) C
* At least 1 year post injury

Exclusion Criteria:

* Spinal cord injuries of other severities (classified ASIA A, B, D, or E)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36
Dates: Start 1998-05; Study Completion 2002-04

CONTACTS AND LOCATIONS:
Overall Officials: Edelle Carmen Field, Ph.D., P.T., Principal Investigator — University of Miami
Locations (1):
- Miami Project, Bantle Center, Miami, Florida, United States

REFERENCES:
- See also: Click here for more information about the Miami Project to Cure Paralysis. — http://www.miamiproject.miami.edu/